CLINICAL TRIAL: NCT04351334
Title: Patient Profiles and Treatment Patterns Among ALK-positive NSCLC Patients Treated With Alectinib
Brief Title: Anaplastic Lymphoma Kinase (ALK)-Positive Non-small Cell Lung Cancer (NSCLC) Post-alectinib Treatment Patterns
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B7461031
Record Dates: First submitted 2020-04-15; First posted 2020-04-17 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-05

CONDITIONS: Non-Small-Cell Lung Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — alectinib

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Patients with ALK-positive NSCLC
  Interventions: Drug: Alectinib

INTERVENTIONS:
Drug: Alectinib — Observational treatment based on physician choice

SUMMARY:
This study aims to understand patient profiles, treatment patterns, and clinical outcomes among ALK-positive NSCLC patients treated with alectinib, and post-alectinib treatment patterns and outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a documented diagnosis of NSCLC.
2. Patients ≥ 18 years of age at initial recorded diagnosis of NSCLC.
3. Patients who received treatment with alectinib during the study identification period, including those who initiated alectinib prior (index date-1) to the start of the study identification period.
4. During the study observation period, patients observed with at least 2 visits after the index date-1.

Exclusion Criteria:

1. Receipt of treatment indicated for another primary cancer or diagnosis of another primary cancer (with the exception of non-melanotic skin cancer), within 5 years of index date-1 will be excluded.
2. Patients enrolled in clinical trials prior to receiving alectinib during the study ID period (index date-1), will be included and flagged in the analysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of patients with a diagnosis of NSCLC receiving alectinib.
Sampling Method: Non-Probability Sample
Enrollment: 161 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Inc, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7461031

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants with anaplastic lymphoma kinase + non-small cell lung cancer (ALK+ NSCLC) who were on treatment with Alectinib during 01 June 2017 and 31 August 2020 were eligible for this study. Data of eligible participants from 01 June 2017 to 31 August 2021, were extracted from iKnowMed (iKM) electronic health record (EHR). Data was evaluated per objectives of this retrospective observational study from 27 March 2020 to 01 November 2022.
Groups:
- All Eligible Participants: Participants who were on treatment with Alectinib for ALK+ NSCLC in real world clinical practices during 01-Jun-2017 to 31-Aug-2020.
Period: Overall Study
Arm/Group | All Eligible Participants
Started | 161
Completed | 161
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Analysis population included all eligible participants whose data were included and observed in this study.
Arm/Group | All Eligible Participants
Number analyzed (Participants) | 161
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.4 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91
  Male | 70
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 10
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 13
  White | 111
  More than one race | 0
  Unknown or Not Reported | 27
Number of Participants According to Practice Region [Count of Participants; unit: Participants] — Number of participants classified according to practice region were reported in this baseline characteristic.
  Participants
    Midwest | 34
    Northeast | 9
    South | 58
    West | 60
Number of Participants Classified According to Smoking History [Count of Participants; unit: Participants] — Number for participants classified according to smoking history were reported in this baseline characteristic.
  Participants
    Current | 5
    Former | 51
    Never | 81
    No information | 24
Number of Participants According to Eastern Cooperative Oncology Group (ECOG) Performance Score [Count of Participants; unit: Participants] — The ECOG performance status score is a rating of a participant's disease status, daily living activities and quality of life, where 0 indicates fully active,1 indicates restricted in physically strenuous activity, 2 indicates ambulatory and capable of self-care but unable to work, 3 indicates capable only of limited self-care, 4 indicates completely disabled and 5 indicates dead. Higher scores indicated more severe disease, difficulty in performing daily activity and poor quality of life.
  Participants
    0 | 18
    1 | 70
    2 | 20
    Greater than or equal to (>=) 3 | 2
    Not documented | 51
Number of Participants According to Tumor Histology [Count of Participants; unit: Participants] — Number of participants classified according to tumor histology were reported in this baseline characteristic.
  Participants
    Adenosquamous carcinoma | 2
    Large cell carcinoma | 1
    Adenocarcinoma | 132
    Other | 2
    Squamous cell carcinoma | 2
    Not documented | 22
Number of Participants According to Stage at Initial NSCLC Diagnosis [Count of Participants; unit: Participants] — In this baseline measure disease stage at initial NSCLC diagnosis was categorized as a) Early stage ((IA, IB, IIA, IIIB, II not specified); b) participants identified as stage III but without any record of A, B or C (III not specified); c) Limited/Regional (IIIA); d) Locally advanced (IIIB, IIIC); e) Metastatic (IV) and f) Unknown. The higher the stage number, the larger the tumor and/or the more it has spread into nearby tissues.
  Participants
    Early Stage (IA, IB, II [not specified], IIA) | 13
    Stage III (Not specified) | 1
    Limited/Regional (IIIA) | 12
    Locally advanced (IIIB/IIIC) | 6
    Metastatic (IV) | 129
Number of Participants According to ROS Proto-Oncogene 1 (ROS1) Status [Count of Participants; unit: Participants] — Number of participants classified according to ROS1 status was reported in this baseline characteristic. Unknown might have included results classified as unknown or pending. Not documented indicated that there was no documentation of testing results.
  Participants
    Positive | 0
    Negative | 78
    Unknown | 15
    Not documented | 68
Number of Participants According to Epidermal Growth Factor Receptor (EGFR) Mutation Status [Count of Participants; unit: Participants] — Number of participants classified according to EGFR mutation status was reported in this baseline characteristic. Unknown might have included results classified as unknown or pending. Not documented indicated that there was no documentation of testing results.
  Participants
    Positive | 2
    Negative | 114
    Unknown | 4
    Not documented | 41
Number of Participants According to v-raf Murine Sarcoma Viral Oncogene Homolog B1 Mutation Status [Count of Participants; unit: Participants] — Number of participants classified according to v-raf murine sarcoma viral oncogene homolog B1 (BRAF) mutation status was reported in this baseline characteristic. Unknown might have included results classified as unknown or pending. Not documented indicated that there was no documentation of testing results.
  Participants
    Positive | 0
    Wild-type | 65
    Unknown | 36
    Not documented | 60
Number of Participants According to Programmed Death-Ligand 1 (PD-L1) Expression [Count of Participants; unit: Participants] — Number of participants classified according to PD-L1 expression was reported in this baseline characteristic. Unknown might have included results classified as unknown or pending. Not documented indicated that there was no documentation of testing results.
  Participants
    1-49 percent (%) Expression | 38
    >= 50% Expression | 38
    Negative | 15
    Unknown | 28
    Not documented | 42

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Classified According to Treatments Received for Anaplastic Lymphoma Kinase Positive-non-Small Cell Lung Cancer (ALK + NSCLC) in Sequence
Description: Number of participants classified according to ALK-TKI treatment patterns or sequencing were reported in this outcome measure.
Time Frame: During the inclusion period from 01-Jun-2017 to 31-Aug-2020 (maximum up to 39 months); eligible data was studied during approximately 31 months of this retrospective study
Population: Analysis population included all eligible participants whose data were included and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | All Eligible Participants
Number analyzed (Participants) | 161
Participants
  Alectinib only | 103
  Alectinib followed by chemotherapy | 8
  Alectinib followed by lorlatinib | 23
  Alectinib followed by crizotinib | 1
  Alectinib followed by immunotherapy | 2
  Alectinib followed by brigatinib | 15
  Alectinib followed by chemoimmunotherapy | 4
  Alectinib followed by ceritinib | 2
  Alectinib followed other | 3

2. Primary Outcome: Number of Participants Classified According to Reason for Alectinib Treatment Discontinuation
Description: Number of participants classified according to reason for Alectinib treatment discontinuation were reported in this outcome measure. One participant could have more than one reason for discontinuation.
Time Frame: From initiation of index treatment to discontinuation from 01-Jun-2017 to 31-Aug-2021 (maximum up to 51 months); eligible data was studied during approximately 31 months of this retrospective study
Population: Analysis population included all eligible participants whose data were included and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | All Eligible Participants
Number analyzed (Participants) | 161
Participants
  Hospice | 7
  Toxicity | 13
  Death | 15
  Progression | 55
  Decline in performance status | 1
  Participant choice | 1
  Physician choice | 1
  Unknown | 3
  Other | 3
  No evidence of alectinib discontinuation | 68

3. Primary Outcome: Duration of Therapy (DOT)
Description: DOT was defined as duration of time between alectinib or post-alectinib treatment initiation and discontinuation as documented in the iKM EHR database. Participants who did not have evidence of discontinuation, starting new therapy, or whose last prescription date was less than (<) 30 days from the end of the study period, were censored at last visit date or end of study period.
Time Frame: Alectinib or post-alectinib treatment initiation till its discontinuation or censoring date, during study observation period (maximum up to 51 months); eligible data was studied during approximately 31 months of this retrospective study
Population: Analysis population included all eligible participants whose data were included and observed in this study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | All Eligible Participants
Number analyzed (Participants) | 161
Months | 23.9 [18.2 to 31.9]

4. Primary Outcome: Overall Survival (OS)
Description: OS was defined as the interval between treatment and the date of death (any cause) as documented in the iKM EHR database. Participants who did not die within the study observation period were censored on the study end date or the last visit date available in the dataset, whichever occurred first.
Time Frame: From start of treatment until date of death or censoring date, during study observation period (maximum up to 51 months); eligible data was studied during approximately 31 months of this retrospective study
Population: Analysis population included all eligible participants whose data were included and observed in this study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | All Eligible Participants
Number analyzed (Participants) | 161
Months | 46.3 [36.6 to NA] — Upper limit of 95% CI could not be estimated as there were insufficient number of participants with event and hence not available to report.

5. Primary Outcome: Progression Free Survival (PFS)
Description: PFS was measured from the initiation of the treatment to the date of progression (documented by provider as disease has progressed or worsening of disease) or date of death due to any cause, censoring participants who were still alive at the end of the study observation period and did not progress at the last visit date.
Time Frame: From initiation of index treatment to date of progression or death due to any cause or censoring date, during study observation period (maximum up to 51 months); eligible data was studied during approximately 31 months of this retrospective study
Population: Analysis population included all eligible participants whose data were included and observed in this study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | All Eligible Participants
Number analyzed (Participants) | 161
Months | 41.4 [20.1 to NA] — Upper limit of 95% CI could not be estimated as there were insufficient number of participants with event and hence not available to report.

ADVERSE EVENTS:
Time Frame: For all-cause mortality: from start of treatment until date of death or censoring date, during study observation period (maximum up to 51 months); eligible data was studied during approximately 31 months of this retrospective study
Description: This observational retrospective study retrieved data from medical records and the data existed as unstructured data. In these data sources, individual participant data were not retrieved or validated, and it was not possible to link a particular product and medical event for any individual. Thus, minimum criteria (identifiable participant, identifiable reporter, a suspect product, and event) for reporting an adverse event could not be met, hence safety data not collected and reported.
Arm/Group | All Eligible Participants
All-Cause Mortality (participants affected / at risk) | 56/161
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-31): https://cdn.clinicaltrials.gov/large-docs/34/NCT04351334/Prot_SAP_000.pdf